CLINICAL TRIAL: NCT06223243
Title: The Effect of Stingless Bee Honey Mouthrinse on Dental Plaque Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Islam Malaysia (Other)
Responsible Party: Principal Investigator, NUR AYMAN ABDUL HAYEI, Clinical Lecturer, Universiti Sains Islam Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SBH Mouthrinse
Record Dates: First submitted 2023-02-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Plaque Accumulation; Patient Acceptance

STUDY DESIGN:
Intervention Model Description: randomised clinical trial, blinded and performed in 3 parallel groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Tthe assessor was not involved in the mouthrinse assignment. Besides, the bottles were covered to prevent from showing the color of mouthrinse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- stingless bee honey (Experimental): stingless bee honey mouthrinse was prescribed to participants assigned to this group.
  Interventions: Other: Stingless bee honey mouthrinse
- chlorhexidine (Active Comparator): chlorhexidine mouthrinse was prescribed to participants assigned to this group.
  Interventions: Other: chlorhexidine mouthrinse
- normal saline (Placebo Comparator): Normal saline mouthrinse was prescribed to participants assigned to this group.
  Interventions: Other: normal saline mouthrinse

INTERVENTIONS:
Other: Stingless bee honey mouthrinse — Three bottles of 90ml of stingless bee honey of 20% concentration was given to each subject. This mouthrinse preparation was instructed for subjects to be taken 30ml each, thrice daily for three days.
  Arms: stingless bee honey
Other: normal saline mouthrinse — Subjects were instructed to rinse with 30ml of normal saline (0.9% concentration) thrice daily for three days.
  Arms: normal saline
Other: chlorhexidine mouthrinse — Subjects were instructed to rinse with 30ml of chlorhexidine mouthrinse thrice daily for three days.
  Arms: chlorhexidine

SUMMARY:
Mouthrinses are recommended as a complement to mechanical methods in oral hygiene procedures to prevent and control periodontal diseases. Chlorhexidine mouthrinse has been used as a chemical plaque control agent for many years. However, in spite of its potent antimicrobial and antiplaque properties, there have been various reports of the undesirable adverse effects of chlorhexidine mouthrinse. This creates the need to look for an alternative mouthrinse that can also help in controlling plaque.

Stingless bee honey is an alternative agent which is increasingly known for its better properties and easily available compared to other types of honey. It has been reported to have many benefits for the oral cavity such as antibacterial, anti-inflammatory, and healing properties which makes it a potential therapeutic agent in periodontal therapy. However, there is a lack of clinical studies showing its efficacy in plaque control as a mouthrinse.

Hence, this study aims to investigate the ability of stingless bee honey mouthrinse to reduce plaque accumulation. This will be done through a randomised clinical trial whereby subjects will be prescribed with a mouthrinse formulation and instructed to refrain from any tooth cleaning procedure. The patient's plaque score will be recorded before and after the intervention to measure the effectiveness of the mouthrinse.

DETAILED DESCRIPTION:
Objectives:

i. To investigate the patients' plaque level after use of stingless bee honey mouthrinse in a clinical trial. ii. To investigate patients' acceptance to stingless bee honey mouthrinse. iii. To compare plaque level after use of stingless bee honey mouthrinse to chlorhexidine mouthrinse.

This is a randomised, double-blinded, placebo-controlled clinical study that will be conducted at the Faculty of Dentistry, Universiti Sains Islam Malaysia (USIM). Application of ethical approval will be made to USIM's medical ethical committee of the Faculty of Medicine and Health Science.

Patients who seek scaling and polishing treatment at Faculty of Dentistry, USIM were invited to participate in study. Written and informed consent were obtained from the participants. As this is a pilot study, sample size calculation was not performed. A total of ten participants per group were recruited for the study.

Pre-intervention, plaque score and BPE were taken at baseline by a single clinician (NAH), a periodontist. This was to reduce any variation in plaque score recording between different clinicians. Both the patients and the clinician were blinded to the intervention given to reduce bias. After recording the plaque score, scaling and prophylaxis were performed by periodontists (NAH, NHMB & MAS). This was to ensure that all participants start at an equal oral hygiene level and that the score taken after three days will be purely from plaque formation and not from the negligence of oral hygiene.

Three different mouthrinse formulations were prepared for this study: (1) stingless bee honey-based mouthrinse (Bayu kelulut ®) containing honey diluted with distilled water to a concentration of 1:1, (2) 0.12% chlorhexidine (Oradex Antibacterial Mouthwash, Malaysia. Reg no: MAL06011901XCZ), and (3) placebo (negative control) containing saline solution. The Malaysian stingless bee honey, Bayu Kelulut ® is a product certified by Malaysian Good Manufacturing Practices and Malaysian Agricultural Research and Development Institute (MARDI), and chlorhexidine is registered under the National Pharmaceutical Regulatory Agency, Ministry of Health. These mouthrinse preparations were packed, sealed and coded in identical bottles before starting the study.

60ml of mouthrinse in a sealed bottle were prescribed by two dental students at random. These formulations were mixed in Laboratory level 18, Faculty of Dentistry, Universiti Sains Islam Malaysia and kept in the refrigerator between 2-8°C. Patients were instructed to refrain from all forms of tooth cleaning and rinse 10ml of mouthrinse twice daily for two minutes. This was done in three days.

After three days, the same clinician (NAH) measured the plaque score and BPE again. Prophylaxis were given.

ELIGIBILITY:
Inclusion Criteria:

1. Medically healthy participants aged between 18-40
2. Healthy gingiva or localised gingivitis with the highest Basic Periodontal Examination (BPE) score of 2
3. Presence of at least 20 natural teeth

Exclusion Criteria:

1. Diabetes
2. Physical and/or mental disabilities that may interfere with receiving mouthrinse instructions
3. Orthodontic or prosthodontic appliances
4. Undergoing antibiotic/antimicrobial therapy
5. Current smoker
6. Abnormal saliva secretion rate
7. Pregnancy
8. Allergy to honey or bee stings

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
plaque score | three days
  plaque accumulation level will be measured using dichotomous scoring system ( 1- presence of plaque and 0- absence of plaque) for each 4 sites in each tooth. The scoring will be added and divided by total number of sites, and results in a percentage (plaque score).

SECONDARY OUTCOMES:
patients' acceptance | 3 days
  patients' acceptance on mouthrinse in terms of halitosis, taste, odour and burning sensation were recorded using visual analogue scale whereby 1 indicates worst experience while 10 indicates best experience.

CONTACTS AND LOCATIONS:
Overall Officials: NUR AYMAN ABDUL HAYEI, Principal Investigator — FACULTY OF DENTISTRY, UNIVERSITI SAINS ISLAM MALAYSIA
Locations (1):
- Students Dental Clinic, Faculty of Dentistry, University Sains Islam Malaysia., Kuala Lumpur, Pandan Indah, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The IPD might be shared if it would expand the results of the study.
Supporting Information: Study Protocol
Time Frame: Two years